CLINICAL TRIAL: NCT04668794
Title: Carpometacarpal Fracture-dislocation of the Hand: Interobserver and Intraobserver Variability for Identify Associate Hamate Fractures and Its Implications in Surgical Planning and Treatment
Brief Title: Carpometacarpal Fracture-dislocations
Acronym: Dislocation
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FLC-2020-29
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Carpometacarpal; Dislocation
MeSH Terms: conditions — Joint Dislocations | interventions — Fracture Fixation, Internal; POLR1G protein, human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Osteosynthesis — Reduction and fixation of the carpometacarpal fracture dislocation of the hand with osteosynthesis (Kirschners wires, plate and screws)
  Other Names: Cast

SUMMARY:
Fracture-dislocation of the carpometacarpal (CMC) joints of the ring and little finger are the most affected CMC joints and the dislocation may be accompanied by other hand injuries. Fracture-dislocation of the CMC joints of the ring and little finger are extremely mobile because of their saddle shape anatomy and loose ligamentous attachments. Missed and incorrect diagnosis is very frequent in metacarpal base injuries of the hand and results in impaired function and weak grip. In these lesions immediate reduction is imperative. Treatment options for these injuries include non-operative management, closed reduction with Kirschner wire fixation (K-wire) and open reduction with internal fixation (ORIF). In chronic CMC fracture-dislocations ORIF is mandatory. Although operative treatment is recommended in the literature in fracture-dislocation of the CMC joints of the ring and little finger, other authors, in specific cases, performed conservative treatment through immediate reduction and splint immobilization and this treatment can be sufficient.

DETAILED DESCRIPTION:
Physical examination in carpometacarpal injuries reveals ulnar-sided pain, swelling, diffuse edema, a palpable lump and tenderness of the hand.

Radiological examination include hand-wrist radiographs in the posteroanterior (PA), true lateral and 45º oblique views. A true lateral view of the hand may demonstrate the dislocation, although overlapping of the joints can mask the dislocation. On PA radiographs, Fisher et al. propose using the so-called M-line parallelism of the CMC joints. A break in this M-line suggests a dislocation. Another method is to draw metacarpal cascade lines on a PA radiographs.

It is important to recognise the associate lesions, for example hamate fractures, because this fracture can change the prognosis, surgical planning and treatment. The investigators hypothesized that there is an interobserver variability to evaluate the carpometacarpal fracture-dislocation and associated lesions in x-rays are underestimated. The investigators propose a protocol with a CT scan to asses this lesions. The researchers hypothesised that surgical reconstruction would result in better clinical result and lower complications rate than non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Closed carpometacarpal fracture dislocation of the hand
* Adults from 18 to 80 years old

Exclusion Criteria:

* history of fractures or tendon lesions in the same hand
* Children
* Open fracture dislocations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are adults with a closed injury in their hand. For clinical, x-ray and TC we evaluated the carpometacarpal fracture dislocation of the hand and associated lesions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Hamate fracture | 6 months
  Hamate fracture associated with the dislocation of the fifth and fourth finger. Cain´s classification for the description of fracture-dislocation. Milch´s classification for hamate fractures types.
Degree of displacement | 6 months
  Degree of displacement (% displacement) in X-rays and CT scan.
Intrarticular stepoff and degenerative osteoarthritis | 6 months
  Intrarticular stepoff (mm) and sclerosis, cysts, osteophytes, joint space reduction (mm) in X-rays and CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Retrospective study that observe the x-rays and TC scan and the results of the surgical or conservative treatment.

REFERENCES:
- [Result] Kural C, Basaran SH, Ercin E, Bayrak A, Bilgili MG, Baca E. Fourth and fifth carpometacarpal fracture dislocations. Acta Orthop Traumatol Turc. 2014;48(6):655-60. doi: 10.3944/AOTT.2014.14.0040. PMID 25637730
- [Result] Gehrmann SV, Kaufmann RA, Grassmann JP, Logters T, Schadel-Hopfner M, Hakimi M, Windolf J. Fracture-dislocations of the carpometacarpal joints of the ring and little finger. J Hand Surg Eur Vol. 2015 Jan;40(1):84-7. doi: 10.1177/1753193414562706. PMID 25538072
- [Result] Mueller JJ. Carpometacarpal dislocations: report of five cases and review of the literature. J Hand Surg Am. 1986 Mar;11(2):184-8. doi: 10.1016/s0363-5023(86)80048-x. PMID 3958446
- [Result] Henderson JJ, Arafa MA. Carpometacarpal dislocation. An easily missed diagnosis. J Bone Joint Surg Br. 1987 Mar;69(2):212-4. doi: 10.1302/0301-620X.69B2.3818751.
- [Result] Kjaer-Petersen K, Jurik AG, Petersen LK. Intra-articular fractures at the base of the fifth metacarpal. A clinical and radiographical study of 64 cases. J Hand Surg Br. 1992 Apr;17(2):144-7. doi: 10.1016/0266-7681(92)90075-d. PMID 1588193
- [Result] Cobb WA, Dingle L, Zarb Adami R, Rodrigues J. Management of fracture-dislocations of the little finger carpometacarpal joint: a systematic review. J Hand Surg Eur Vol. 2018 Jun;43(5):530-538. doi: 10.1177/1753193417752317. Epub 2018 Feb 7. PMID 29411672
- [Result] Storken G, Bogie R, Jansen EJ. Acute ulnar carpometacarpal dislocations. Can it be treated conservatively? A review of four cases. Hand (N Y). 2011 Dec;6(4):420-3. doi: 10.1007/s11552-011-9347-3. Epub 2011 Jul 7. No abstract available. PMID 23204970
- [Result] Fisher MR, Rogers LF, Hendrix RW. Systematic approach to identifying fourth and fifth carpometacarpal joint dislocations. AJR Am J Roentgenol. 1983 Feb;140(2):319-24. doi: 10.2214/ajr.140.2.319. PMID 6600352
- [Result] Hodgson PD, Shewring DJ. The 'metacarpal cascade lines'; use in the diagnosis of dislocations of the carpometacarpal joints. J Hand Surg Eur Vol. 2007 Jun;32(3):277-81. doi: 10.1016/J.JHSB.2006.09.020. PMID 17331628
- [Derived] Fa-Binefa M, Almenara M, Mata-Munoz JM, Gich-Saladich I, Llauger J, Lamas C. Retrospective interobserver agreement on diagnoses of 4th and 5th carpometacarpal fracture-dislocation and hamate fracture in plain X-ray - Is CT essential after ulnar carpometacarpal pain? Skeletal Radiol. 2023 Dec;52(12):2427-2433. doi: 10.1007/s00256-023-04366-9. Epub 2023 May 25. PMID 37227483